CLINICAL TRIAL: NCT02728934
Title: Comparative and Pragmatic Study of Simponi Aria Versus Remicade in Rheumatoid Arthritis
Brief Title: Comparative and Pragmatic Study of Golimumab Intravenous (IV) (Simponi Aria) Versus Infliximab (Remicade) in Rheumatoid Arthritis
Acronym: AWARE
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108132; CNTO148ART4011 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Golimumab; Infliximab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab; Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Golimumab Intravenous (IV): Patients in the US who enroll in the study will have a rheumatologist confirmed diagnosis of Rheumatoid arthritis (RA) and will be medically eligible for, and will have been prescribed but not yet initiated treatment with Golimumab IV.
  Interventions: Biological: Golimumab Intravenous (IV)
- Infliximab: Patients in the US who enroll in the study will have a rheumatologist confirmed diagnosis of Rheumatoid arthritis (RA) and will be medically eligible for, and will have been prescribed but not yet initiated treatment with Infliximab.
  Interventions: Biological: Infliximab; Biological: Biosimilar Infliximab

INTERVENTIONS:
Biological: Golimumab Intravenous (IV) — This is an observational study. Patients who will receive golimumab IV will be observed for 3 years.
  Other Names: Simponi Aria
  Groups: Golimumab Intravenous (IV)
Biological: Infliximab — This is an observational study. Patients who will receive infliximab will be observed for 3 years.
  Other Names: Remicade
  Groups: Infliximab
Biological: Biosimilar Infliximab — This is an observational study. New patients who will receive biosimilar infliximab will be observed for 3 years (maximum). Biosimilar Infliximab patients will be included in Exploratory analyses only and will not be included in Primary or Secondary outcome measures analyses.
  Other Names: Inflectra
  Groups: Infliximab

SUMMARY:
The purpose of this study is to compare the proportion of patients with an infusion reaction in Rheumatoid arthritis (RA) patients treated with Golimumab Intravenous (IV) or Infliximab.

DETAILED DESCRIPTION:
This is a prospective, noninterventional (no treatment medication provided by the study), observational (study in which the investigators/ physicians observe the patients and measure their outcomes), multicenter (study conducted at multiple sites) study of Golimumab IV and Infliximab in RA patients. The study allows for an anticipated 2-year enrollment period and a 3-year study duration for each patient. No interventions will be given to patients as a part of this study. This study will be conducted in the US, at rheumatology-based clinical practices and will enroll adult RA patients who meet all entry criteria. The primary endpoint of this study is the proportion of patients with an infusion reaction through week 52. Patients will be enrolled in a 1:1 ratio to initiate treatment with either Golimumab IV or Infliximab. Patients' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be a male or female 18 years of age or older as the study is intended to assess Golimumab intravenous (IV) and Infliximab in adult RA patients
* Patient must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study
* Patient has a confirmed diagnosis of Rheumatoid arthritis (RA) and is medically eligible for treatment with Golimumab IV or Infliximab in accordance with standard of care (example, screening for tuberculosis [TB], vaccinations, etc.)
* At the time of enrollment the patient will be initiating treatment with Golimumab IV or Infliximab. The patient may or may not have previously received treatment with a biologic. Patients with previous exposure to subcutaneously administered Simponi may enroll in the study
* Patient must be willing to complete Patient reported outcomes (PRO) forms during the study and agree to return completed forms to the site if receiving an infusion of Golimumab IV or Infliximab at a location remote from the study site

Exclusion Criteria:

* Patient is less than 18 years of age
* Patient is pregnant or planning a pregnancy
* Patient is currently enrolled in an interventional study
* Patient has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 28 days, as appropriate, before the planned first dose of Golimumab IV or Infliximab
* Patient previously received Golimumab IV if planning to receive Golimumab IV in this study or the patient previously received Infliximab if planning to receive Infliximab or BI in this study. Patient previously receive BI if planning to receive BI or Remicade in this study
* Patient has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (example, compromise the patient's well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the US who enroll in the study will have a rheumatologist confirmed diagnosis of Rheumatoid arthritis (RA) and will be medically eligible for, and will have been prescribed but not yet initiated treatment with, either Golimumab IV or Infliximab.
Sampling Method: Non-Probability Sample
Enrollment: 1279 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients With an Infusion Reaction Through Week 52 | Up to week 52
  An infusion reaction is any adverse event that occurs during an infusion or within 1 hour of completion of infusion of either Golimumab IV or Infliximab. The number of patients with infusion reactions will be reported.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Disease Activity Index (CDAI) Score in Bionaïve Patients at Month 6 | Baseline and Month 6
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. The change from baseline at Month 6 in CDAI in bionaive patients will be reported.
Change from Baseline in CDAI Score in Bionaïve Patients at Month 12 | Baseline and Month 12
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. The change from baseline at Month 12 in CDAI in bionaïve patients will be reported.
Change from Baseline in CDAI Score in Bionaïve Patients at Month 3 | Baseline and Month 3
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. The change from baseline at Month 3 in CDAI in bionaïve patients will be reported.
CDAI Score in Patients with or Without Concomitant Methotrexate use | Months 3, 6, 12, and at 6-month intervals through the end of the study (up to Month 36)
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. CDAI score in patients with or without concomitant methotrexate use, will be reported.
Change from Baseline in CDAI Score in Patients with or Without Concomitant Methotrexate use | Baseline, Months 3, 6, 12, and at 6-month intervals through the end of the study (up to Month 36)
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. Change from baseline in CDAI score in patients with or without concomitant methotrexate use, will be reported.
CDAI Score in Dose-escalated Patients | Months 6, 12, and at 6-month intervals through the end of the study (up to Month 36)
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. CDAI score in patients in whom dose of Remicade was escalated (increased prescribe dose or reduced dose interval, or a combination of both), will be reported.
Change from Baseline in CDAI Score in Dose-escalated Patients | Baseline, Months 6, 12, and at 6-month intervals through the end of the study (up to Month 36)
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. Change from baseline in CDAI score in patients in whom dose of Remicade was escalated (increased prescribe dose or reduced dose interval, or a combination of both), will be reported.
CDAI Score in Patients who Previously Administered Remicade (or Other Biologic[s]) | Months 3, 6, 12, and at 6-month intervals through the end of the study (up to Month 36)
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. CDAI score in patients who previously administered Remicade (or other biologic[s]), will be reported.
Change from Baseline in CDAI Score in Patients who Previously Administered Remicade (or Other Biologic[s]) | Baseline, Months 3, 6, 12, and at 6-month intervals through the end of the study (up to Month 36)
  The CDAI is a validated measure of disease activity consisting of the sum of 4 clinical variables: tender joint and swollen joint count based on a 28-joint assessment, patient global assessment, and the physician global assessment of disease activity based on a visual analog scale (VAS) ranging from 0 to 10. The CDAI has a range from 0 to 76, with higher scores indicating more severe disease. Change from baseline in CDAI score in patients who previously administered Remicade (or other biologic[s]), will be reported.
Number of Patients With Serious Infusion Reaction and Discontinuation of Therapy due to Infusion Reaction | 3 years
Number of Infusions With Infusion Reactions | 3 years
Discontinuation Rates | 3 years
  Participants discontinuation rates for both the Simponi Aria and Remicade groups will be reported.
Persistency of use of Treatment | 3 years
  Persistency of use, defined as the continuous period of time a participant receives either Simponi Aria or Remicade, will be reported.
Number of Patients with Adverse Events (AEs) and Serious AEs | 3 years
Number of Patients With an Infusion Reaction | 3 years
Number of Patients With Severe Infusion Reaction and Discontinuation of Therapy due to Infusion Reaction | Up to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (85):
- United States (85):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Prescott, Arizona
  - Sun City, Arizona
  - Bakersfield, California
  - Campbell, California
  - Covina, California
  - El Cajon, California
  - Hemet, California
  - Los Angeles, California
  - Santa Cruz, California
  - Thousand Oaks, California
  - Upland, California
  - Van Nuys, California
  - West Hills, California
  - Whittier, California
  - Denver, Colorado
  - Lakewood, Colorado
  - Clearwater, Florida
  - Palm Harbor, Florida
  - Plantation, Florida
  - Tamarac, Florida
  - Venice, Florida
  - Lawrenceville, Georgia
  - Springfield, Illinois
  - Muncie, Indiana
  - Bowling Green, Kentucky
  - Baton Rouge, Louisiana
  - Monroe, Louisiana
  - Shreveport, Louisiana
  - Cumberland, Maryland
  - Hagerstown, Maryland
  - Towson, Maryland
  - Wheaton, Maryland
  - Ann Arbor, Michigan
  - Lansing, Michigan
  - Saint Clair Shores, Michigan
  - Eagan, Minnesota
  - Edina, Minnesota
  - Las Vegas, Nevada
  - Nashua, New Hampshire
  - Freehold, New Jersey
  - Voorhees Township, New Jersey
  - Brooklyn, New York
  - Orchard Park, New York
  - Greensboro, North Carolina
  - Leland, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Edmond, Oklahoma
  - Tulsa, Oklahoma
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wexford, Pennsylvania
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Amarillo, Texas
  - Beaumont, Texas
  - College Station, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Mesquite, Texas
  - Nassau Bay, Texas
  - Plano, Texas
  - San Antonio, Texas
  - San Marcos, Texas
  - Sugar Land, Texas
  - The Woodlands, Texas
  - Waco, Texas
  - Arlington, Virginia
  - Chesapeake, Virginia
  - Newport News, Virginia
  - Kennewick, Washington
  - Seattle, Washington
  - Beckley, West Virginia
  - South Charleston, West Virginia
  - Glendale, Wisconsin
  - Onalaska, Wisconsin

REFERENCES:
- [Derived] Broadwell A, Schechtman J, Conaway D, Kivitz A, Shiff NJ, Black S, Xu S, Langholff W, Schwartzman S, Curtis JR. Effectiveness and safety of intravenous golimumab with and without concomitant methotrexate in patients with rheumatoid arthritis in the prospective, noninterventional AWARE study. BMC Rheumatol. 2023 Mar 27;7(1):5. doi: 10.1186/s41927-023-00329-8. PMID 36973741
- [Derived] Bingham CO 3rd, Black S, Shiff NJ, Xu S, Langholff W, Curtis JR. Response to Treatment with Intravenous Golimumab or Infliximab in Rheumatoid Arthritis Patients: PROMIS Results from the Real-World Observational Phase 4 AWARE Study. Rheumatol Ther. 2023 Jun;10(3):659-678. doi: 10.1007/s40744-023-00533-5. Epub 2023 Feb 23. PMID 36820983
- [Derived] Curtis JR, Chakravarty SD, Black S, Kafka S, Xu S, Langholff W, Parenti D, Greenspan A, Schwartzman S. Incidence of Infusion Reactions and Clinical Effectiveness of Intravenous Golimumab Versus Infliximab in Patients with Rheumatoid Arthritis: The Real-World AWARE Study. Rheumatol Ther. 2021 Dec;8(4):1551-1563. doi: 10.1007/s40744-021-00354-4. Epub 2021 Aug 20. PMID 34417735